CLINICAL TRIAL: NCT05710354
Title: Russian Multicenter Comparative Low-intervention Study of the Impact of Perioperative High-protein Nutritional Support on Postoperative Outcomes in the Treatment of Primary Lung Cancer
Brief Title: The Study of High-protein Nutritional Support Impact on Postoperative Outcomes in Patients With Primary Lung Cancer
Status: Completed | Type: Observational
Sponsor: Enrollme.ru, LLC (Network)
Collaborators: Danone Nutricia (Industry)
Responsible Party: Sponsor
Other Study IDs: NUTRILUNC
Record Dates: First submitted 2023-01-24; First posted 2023-02-02 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-02

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- The Study Group: Patients in the study group (N=57), in addition to the usual diet, received nutritional support with the Oral Nutrition Supplement (ONS) Nutridrink Compact Protein in the amount of 2 bottles per day for 14 days prior to surgery and 14 days following surgery. During the hospital stay, additional nutritional support was added to the patient's standard hospital diet. On an outpatient basis, the patient received the required amount of ONS at his/her disposal and took it as a supplement to his/her usual and habitual diet. The ONS was recommended to be taken between main meals
  Interventions: Dietary Supplement: Nutridrink Compact Protein
- The Control Group: Patients in the control group (N=57) followed the standard hospital diet, and at outpatient basis - their usual habitual diet

INTERVENTIONS:
Dietary Supplement: Nutridrink Compact Protein — Oral Nutritional Supplement, a liquid, ready-to-drink, high protein, high calorie blend. Intended for adult patients (from 18 years of age) with malnutrition or risk of its development. Produced by Nutricia
  Groups: The Study Group

SUMMARY:
The study was aimed to evaluate the impact of perioperative nutritional support with high-protein mixtures on the risk of postoperative complications, postoperative recovery of respiratory functions in patients with lung cancer, nutritional status and quality of life of patients. Possible adverse events were also studied and described.

DETAILED DESCRIPTION:
The study enrolled 114 patients with primary non-small cell lung cancer and nutritional deficiencies or at risk of developing them, admitted for surgical treatment and meeting other inclusion/exclusion criteria. Patients were randomly divided into two groups: the study group of 57 people and the control group of 57 people.

Patients in the study group, in addition to the usual diet, received nutritional support. During the hospital stay, additional nutritional support was added to the patient's standard hospital diet. On an outpatient basis, patients received the required amount at their disposal and will take it as a supplement to his usual and habitual diet.

Patients in the control group followed the standard hospital diet, and at discharge - the usual habitual diet.

The study was conducted using Enrollme.ru electronic platform. In total, the study comprised screening and 5 visits.

ELIGIBILITY:
Inclusion Criteria:

* Presence of morphological verification of non-small cell lung cancer (NSCLC) without distant metastases;
* Appointment of surgical treatment for primary lung cancer with anatomical resection of the lung (lobectomy, bilobectomy or pneumonectomy);
* Nutritional deficiency or risk of its development (≥3 points on the Nutrition Risk Screening 2002 (NRS-2002) scale);
* No history of nutritional support;
* ECOG (Eastern Cooperative Oncology Group Performance Status Scale) score 0 - 2;
* Life expectancy over 3 months;
* Absence of serious diseases of the gastrointestinal tract, disorders of the liver, kidneys, systemic blood diseases and metabolic disorders at the time of inclusion in the study;
* Absence of severe uncontrolled concomitant chronic diseases and acute diseases (including infectious ones);
* Availability of signed informed consent for inclusion in the study and processing of personal data

Exclusion Criteria:

* Terminal state of the patient, ECOG (Eastern Cooperative Oncology Group Performance Status Scale) 3-4;
* State of refractory cachexia;
* Bleeding, serious injury or blood transfusions in the previous 6 months;
* Decay / abscess in the area of the tumor lesion;
* Presence at the same time of a tumor process of another localization, metastatic lesion of the lungs;
* The presence of concomitant diseases in the stage of decompensation;
* Pregnancy or lactation;
* Allergy to or intolerance to any of the components of Nutridrink Compact Protein, galactosemia, allergy to cow's milk proteins;
* The presence of contraindications to the use of enteral nutrition
* Participation in another study currently or in the past 30 days;
* Any other medical or non-medical reason that, in the physician's opinion, may prevent the patient from participating in the study

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary lung cancer patients were enrolled in the study with or at risk of nutritional malnutrition admitted for surgery and meeting the inclusion/non-inclusion
Sampling Method: Non-Probability Sample
Enrollment: 114 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
Weight | during observation up to 6 weeks
  The weight was measured at each visit
Days in hospital | during observation up to 6 weeks
  Count of hospital stay after surgery
Six Minute Walk Test | during observation up to 6 weeks
  A test to count walk distance a patient can afford during 6 minutes
Hand strength | during observation up to 6 weeks
  A hand strength was measured using hand dynamometer at each visit
Lung complications | during hospital stay for about 2 weeks
  Number of lung postoperative complications, e.g. lung infections, atelectasis were registered

SECONDARY OUTCOMES:
Serum total protein | during observation up to 6 weeks
  Serum total protein was measured at each visit
Serum albumin | during observation up to 6 weeks
  Serum albumin was measured at each visit
Total lymphocyte count | during observation up to 6 weeks
  Serum albumin was measured at each visit
EORTC QLQ-C30 | during observation up to 6 weeks
  EORTC QLQ-C30 (The European Organization for Research and Treatment of Cancer core quality of life questionnaire) questionnaire was completed at visits. The questionnaire incorporates five functional scales, three symptom scales, a global health status, and a number of single items assessing additional symptoms commonly reported by cancer patients. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. Thus a high score for a functional scale and global health status represents a high / healthy level of functioning, but a high score for a symptom scale / item represents a high level of symptomatology / problems

CONTACTS AND LOCATIONS:
Overall Officials: Larisa Volf, Dr, Study Director — Danone Nutricia
Locations (4):
- Russia (4):
  - Omsk Clinical Oncology health center, Omsk
  - Mechnikov Medical University, Saint Petersburg
  - Scientific Medical center Institute of Phthisiopulmonology, Saint Petersburg
  - Smolensk region Clinical Oncology health center, Smolensk